CLINICAL TRIAL: NCT00899262
Title: Early Detection of Lung Cancer: Metabolic Biomarkers for High Risk Screening (MEDLUNG)
Brief Title: Biomarkers for Early Detection of Lung Cancer in Patients With Lung Cancer, Participants at High-Risk for Developing Lung Cancer, or Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South West Wales Cancer Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000599372; SWWCI-MEDLUNG; UKCRN-4682; EU-20862
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Lung Cancer; Tobacco Use Disorder
Keywords: lung cancer; tobacco use disorder
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Disorder | interventions — Immunohistochemistry; Spectroscopy, Fourier Transform Infrared

INTERVENTIONS:
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: sputum cytology
Procedure: Fourier transform infrared spectroscopy
Procedure: diagnostic bronchoscopy

SUMMARY:
RATIONALE: Collecting and storing samples of sputum and tissue to study in the laboratory may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking samples of sputum and tissue from lung cancer patients, participants at high risk for developing lung cancer, and from healthy volunteers (both smokers and non-smokers).

DETAILED DESCRIPTION:
OBJECTIVES:

* To test and make a preliminary assessment of the sensitivity and specificity of Fourier transform infrared technology (FTIR) for use in the early detection of lung cancer in sputum samples from patients who have or participants at high risk for developing lung cancer and from non-high-risk smoking and non-smoking volunteers.
* To permit identification of specific metabolic biomarkers within FTIR spectra that can distinguish between lung cancer, high-risk, and non-high-risk cases.

OUTLINE: This is a multicenter study.

Sputum samples and endobronchial biopsy tissue specimens are collected prior to routine bronchoscopy as part of a standard clinical assessment for the early detection of lung cancer. Sputum samples are examined for levels of bronchial and non-bronchial cells using established cytological and immunohistochemical procedures. Samples are also examined for metabolic biomarkers using Fourier transform infrared spectroscopy (FTIR) to generate complete metabolic fingerprints (i.e., spectra) that can distinguish metabolic differences between cancer, non-cancer, and early disease (i.e., dysplasia or metaplasia). These molecular biomarkers, which are detected within FTIR spectra, may be further analyzed in matched endobronchial biopsy tissue samples for histological confirmation. Additional clinico-pathological data is collected for each participant to allow development of predictive statistical models from the data.

All study participants are followed annually.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Diagnosis of lung cancer
  * At high risk for developing lung cancer
  * Non-high-risk smoking or non-smoking volunteer (control)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Development of a cost-effective, high-throughput, and non-invasive screening test using Fourier transform infrared technology for detection of early lung cancer in sputum of high-risk people
Discovery and characterization of novel metabolic biomarkers in sputum samples that permit detection of lung cancer at pre-cancerous and early lung cancer stages

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Lewis, BSc, PhD, Principal Investigator — Swansea University
Locations (2):
- United Kingdom (2):
  - Prince Philip Hospital, Llanelli, Wales
  - South West Wales Cancer Institute, Swansea, Wales

REFERENCES:
- [Result] Lewis PD, Lewis KE, Ghosal R, Bayliss S, Lloyd AJ, Wills J, Godfrey R, Kloer P, Mur LA. Evaluation of FTIR spectroscopy as a diagnostic tool for lung cancer using sputum. BMC Cancer. 2010 Nov 23;10:640. doi: 10.1186/1471-2407-10-640. PMID 21092279